CLINICAL TRIAL: NCT04284683
Title: Physical Activity, Meal Composition, and RMR Among Children Adolescent and Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Dan Nemet, MD, Prof. Dan Nemet, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MeirMc0173-18CTIL
Record Dates: First submitted 2019-03-17; First posted 2020-02-26 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Obesity
Keywords: RMR; Macro nutrients; Exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Proteins; CD36 Antigens; Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal and overweight participants (Experimental): Healthy males and female, age 6 to 30. BMI range for participants age 6 to 18 is between 5th percentile to 85th percentile, overweight BMI between the 85 and 95th percentile, and obese, above the 95th percentile.
  BMI range for participants age 18 to 30 is between 18.5 to 24.9 for normal weight, 25-30 for overweight and above 30 for obese.
  Interventions: Other: DRINK - Water, Protein, Fat, Carbohydrate

INTERVENTIONS:
Other: DRINK - Water, Protein, Fat, Carbohydrate — Following exercise participants will consume a drink (with different composition in each visit) and than RMR will be evaluated.

SUMMARY:
Resting metabolic rate (RMR) is the amount of energy the body uses at rest, and accounts for 60%-70% of daily energy expenditure. Although measured at rest, RMR is strongly influenced by physical activity because the increased metabolic rate during exercise is partially carried over even when exercise stops. Therefore, persons who are physically active maintain higher RMR and less body fat than do sedentary controls. It is well known that high energy intake stimulates whereas caloric restriction reduces RMR. Food thermogenesis corresponds to approximately 10% of daily energy expenditure. Diet-induced thermogenesis is greater on a high protein and carbohydrate diet than on a fat diet. Other factors the affect RMR are age (RMR tends to decline progressively over the life span) and body composition (lean body mass is regarded as the main determinant of RMR). However, the research regarding the effect of a specific combination of macronutrients and exercise on RMR is scarce.

Therefore, the aim of the current study is to assess the combined effect of a meal composition and physical activity on RMR in normal weight and overweight children, adolescents and adults.

DETAILED DESCRIPTION:
One hundred (100) healthy volunteers, 50 normal weight (NW) and 50 overweight (OW), age 6-30 will be recruited for the current study. All participants and/or their parents will sign informed consent prior to their participation. Participants will visit the clinic 4 times, with a week's difference between them. Participants will arrive at the clinic after 12 hours of fasting and avoiding physical activity for 14 hours. During the first visit, their RMR will be measured, and 15min later they will perform 60 min of aerobic training, and 15 minutes later they will be asked to drink 300ml of water, followed by a second RMR test. In the consecutive visits they will follow the same routine without the first RMR test, and drink either carbohydrate enriched shake, protein enriched shake or fat enriched shake; in a random order.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-30 years.
* Normal weight and over weight participants

Exclusion Criteria:

* Elite athletes
* Participants with physical limitations concerning strenuous physical activity.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Change in RMR from baseline | Through study completion, an average of 6 weeks (during 4 visits)
  Resting Metabolic Rate

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - 'Meir children's sport and health center', Kfar Saba
  - Meir Medical Center, Kfar Saba

IPD SHARING:
Plan to Share IPD: No